CLINICAL TRIAL: NCT01302860
Title: A One-year Open-label, Multicenter Trial to Assess Efficacy, Safety and Tolerability of Canakinumab (ACZ885) and the Efficacy and Safety of Childhood Vaccinations in Patients Aged 4 Years or Younger With Cryopyrin Associated Periodic Syndromes (CAPS)
Brief Title: Efficacy, Safety and Tolerability of ACZ885 in Pediatric Patients With the Following Cryopyrin-associated Periodic Syndromes: Familial Cold Autoinflammatory Syndrome, Muckle-Wells Syndrome, or Neonatal Onset Multisystem Inflammatory Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885D2307; 2009-016859-22
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Cryopyrin-associated Periodic Syndromes; Familial Cold Autoinflammatory Syndrome; Muckle-Wells Syndrome; Neonatal Onset Multisystem Inflammatory Disease
Keywords: Cryopyrin-associated periodic syndromes (CAPS); Familial Cold Autoinflammatory Syndrome (FCAS); Muckle-Wells Syndrome (MWS) or Neonatal Onset Multisystem Inflammatory Disease (NOMID); children; systemic autoinflammatory disease; CIAS-1 gene; NALP-3; NLRP3; ACZ885; Ilaris; human monoclonal anti-human interleukin-1 beta (IL-beta); antibody; autosomal dominant; familial autoinflammatory syndrome
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Multiple Pterygium Syndrome, Autosomal Dominant | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Canakinumab (Experimental): Canakinumab s.c. injection (2 mg/kg) was administered every 8 weeks.
  Interventions: Drug: ACZ885

INTERVENTIONS:
Drug: ACZ885

SUMMARY:
This trial will assess the safety, efficacy and tolerability of ACZ885 in patients aged 4 years and younger with cryopyrin associated periodic syndromes (CAPS)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients that are 28 days up to 60 months of age at the time of the screening visit.
2. Body weight > or = 2.5 kg.
3. Parent or legal guardian's written informed consent is required before any assessment is performed for patients.
4. At study entry, patients should have a clinical diagnosis of FCAS, MWS, or NOMID and symptoms requiring pharmacological intervention. Prior agreement between the Investigator and Novartis for study eligibility is required for patients who do not have a molecular diagnosis of NALP3 mutations available (either testing not performed, or testing performed but negative) upon study entry. For those patients who have not been molecularly tested for NALP3 mutations, molecular testing should be performed during the course of the study.
5. For patients treated with an IL-1 blocking agent (i.e. anakinra, rilonacept), these treatments should be discontinued prior to the baseline visit and patients must demonstrate active disease prior to treatment.
6. Patients who are scheduled to receive an immunization, according to their local vaccination guidelines, with an inactivated vaccine must be willing to participate in the assessment schedule for vaccinated patients.

Exclusion Criteria:

1. Preterm neonates for whom, in the Investigator's judgment, participation in the study is not deemed appropriate.
2. History of recurrent and/or evidence of active bacterial, fungal, or viral infections (including HIV).
3. Patients with immunodeficiency or treatment with immunosuppressive drugs.
4. Live vaccinations within < or = 3 months prior to screening. No live vaccinations will be allowed throughout the course of this study and up to 3 months following the last dose.
5. Patients with an increased risk of tuberculosis (TB) infection according to following risk factors:

   * Patients with recent close contact with persons known to have active pulmonary TB disease
   * Foreign-born patients from countries with a high prevalence of tuberculosis
   * Patients with recent tuberculosis infection (including children > 6 months with a positive PPD test [defined as an induration of at least 10mm])
   * Patients with end-stage renal disease
   * Patients with diabetes mellitus
   * Patients receiving immunosuppressive therapy
   * Patients with hematologic cancers.
6. Participation in another trial within the last 30 days or 5 half-lives of the investigational compound (whichever is longer).
7. Familial and social conditions rendering regular medical assessment not possible.
8. Pediatric patients with neutropenia (absolute neutrophil count [ANC] < 1.5 x 10 to the 9th/l)

Other protocol defined inclusion/exclusion criteria may apply

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Laken
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Le Kremlin-Bicêtre, France
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Sankt Augustin
  - Novartis Investigative Site, Tübingen
- Spain (2):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Lausanne, Switzerland
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Brogan PA, Hofer M, Kuemmerle-Deschner JB, Kone-Paut I, Roesler J, Kallinich T, Horneff G, Calvo Penades I, Sevilla-Perez B, Goffin L, Lauwerys BR, Lachmann HJ, Uziel Y, Wei X, Laxer RM. Rapid and Sustained Long-Term Efficacy and Safety of Canakinumab in Patients With Cryopyrin-Associated Periodic Syndrome Ages Five Years and Younger. Arthritis Rheumatol. 2019 Nov;71(11):1955-1963. doi: 10.1002/art.41004. Epub 2019 Sep 9. PMID 31161734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 centers in 7 countries.
Pre-assignment Details: A total of 17 participants were enrolled into the study.
Groups:
- Canakinumab: Participants received body weight stratified dose of canakinumab 2 milligrams/kilogram (mg/kg) subcutaneous (s.c.) injection every 8 weeks.
Period: Overall Study
Arm/Group | Canakinumab
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed in Full analysis set population, defined as all participants who received at least one dose of study drug under this study protocol.
Groups:
- Canakinumab: Participants received body weight stratified dose of canakinumab 2 mg/kg s.c. injection every 8 weeks.
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.9 (1.39)
Age, Customized [Number; unit: participants]
  Infants and toddlers (28 days-23 months) | 6
  Children (2-5 years) | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Aged 4 Years or Younger With at Least One Complete Response at Week 56
Description: Complete response was defined as clinical remission and serological remission. Clinical remission was defined as Physician global assessment of auto-inflammatory disease activity as absent or minimal (using a 5-point scale ranging from absent to severe) and assessment of skin disease as absent or minimal (using a 5-point scale ranging from absent to severe). Serological remission was defined as C reactive protein (CRP) or Serum amyloid A protein (SAA) to be less than (<) 15 milligram per liter (mg/L) and <10 mg/L respectively.
Time Frame: Week 56
Population: The analysis was performed in Full analysis set (FAS), defined as all participants who received at least one dose of study drug under this study protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
Percentage of participants | 94.1

2. Secondary Outcome: Percentage of Participants Aged 2 Years or Younger With at Least One Complete Response at Week 56
Description: Complete response was defined as clinical remission and serological remission. Clinical remission was defined as Physician global assessment of auto-inflammatory disease activity as absent or minimal (using a 5-point scale ranging from absent to severe) and assessment of skin disease as absent or minimal (using a 5-point scale ranging from absent to severe). Serological remission was defined as CRP or SAA to be <15 mg/L and <10 mg/L respectively.
Time Frame: Week 56
Population: The analysis was performed in FAS population. Here, "Number of participants analysed" signifies participants aged 2 years or younger.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 10
Percentage of participants | 90

3. Secondary Outcome: Percentage of Participants With Defined Grades in Physician's Global Assessment Score at Week 56
Description: Participants were assessed based by physician on Physician's Global Assessment measured on a 5--point scale for auto inflammatory disease activity as: 0 = None/absent; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Week 56
Population: The analysis was performed in FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
Percentage of participants
  Absent | 70.6
  Minimal | 23.5
  Mild | 0
  Moderate | 5.9
  Severe | 0

4. Secondary Outcome: Percentage of Participants With Defined Grades in Physician Assessment of Skin Disease at Week 56
Description: Participants were assessed by physician for skin disease (urticarial skin rash) measured on a 5--point scale as: 0 = None/absent; 1 = Minimal; 2 = Mild; 3 = Moderate; 4 = Severe.
Time Frame: Week 56
Population: The analysis was performed in FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
Percentage of participants
  Absent | 82.4
  Minimal | 5.9
  Mild | 11.8
  Moderate | 0
  Severe | 0

5. Secondary Outcome: Change From Baseline in C--Reactive Protein (CRP) and Serum Amyloid A (SAA) Concentrations at Week 56
Description: The CRP and SAA were used as inflammatory markers. The target level concentrations for CRP and SAA was ≤15 mg/L and ≤10 mg/L, respectively. Negative change in concentration of inflammatory markers indicated improvement.
Time Frame: Baseline, Week 56
Population: The analysis was performed in FAS population. Here 'n' signifies those participants with evaluable measurements at both baseline and the post-baseline visit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
mg/L
  CRP (n=14) | -5.4 (6.28)
  SAA (n=16) | -54.4 (133.81)

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: Day 1 (start of study treatment) up to Week 56 (end of study)
Population: The analysis was performed in the safety set population defined as participants who received at least one dose of study drug. Here, 'n' signifies participants evaluable for this measure at specified time points for each group, respectively.
Measure: Number; unit: participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
participants
  AEs (Overall, n=17) | 17
  SAEs (Overall, n=17) | 4
  AEs (Participants <=2 years, n=10) | 10
  SAEs (Participants <=2 years, n=10) | 3

7. Secondary Outcome: Percentage of Participants Receiving a Concomitant Vaccination During the Study
Description: Participants received any one of the following inactivated vaccines as per the immunization program: Corynebacterium diphtheria, Bordetella pertussis, Neisseria meningitidis, Clostridium tetani, Influenza type A, Influenza type B, Haemophilus influenza B, Streptococcus pneumoniae, or Hepatitis B were determined.
Time Frame: Day 1 (start of study treatment) to Week 56 (end of study)
Population: The analysis was performed in the FAS population.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 17
Percentage of participants | 41.2

8. Secondary Outcome: Number of Vaccination Cases With Protective Antibody Levels Following Immunization With Inactivated Vaccines
Description: Participants who received any inactivated vaccines during the study were assessed for their ability to attain protective antibody levels against the vaccine (antigen) post immunization. Participants vaccinations were not assessed for a response if the antibody titre was already sufficient at pre-dose and maintained during the study.
Time Frame: Day -14 (prior-vaccination), Day 0 (vaccination), Day 28, Day 57 (post-vaccination)
Population: The analysis was performed in the FAS population. Here, "Number of participants analysed" signifies evaluable participants who received a total of 31 vaccinations during the study.
Measure: Number; unit: vaccination cases
Arm/Group | Canakinumab
Number analyzed (Participants) | 7
vaccination cases
  Positive response for antibody levels | 18
  No pre-dose antibody levels | 13

9. Secondary Outcome: Number of Participants With Anti-canakinumab Antibodies at Week 56
Description: Immunogenicity assessment included determination of anti-canakinumab (ACZ885) antibodies in serum samples using BIAcore system, with detection based on surface plasmon resonance technique.
Time Frame: Week 56 (End of study)
Population: The analysis was performed in the safety set population. Here, 'Number of participants analysed' signifies participants who had immunogenicity samples taken and analyzed during the study.
Measure: Number; unit: participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 15
participants | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events are monitored from date of First Participant First Visit (FPFV) until Last Participant Last Visit (LPLV), for up to 4 years. All other adverse events are monitored from First Participant First Treatment until LPLV, for up to 4 years.
Arm/Group | Canakinumab
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=17)
Cryopyrin associated periodic syndrome (Congenital, familial and genetic disorders) | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=17)
Eosinophilia (Blood and lymphatic system disorders) | 1
Cryopyrin associated periodic syndrome (Congenital, familial and genetic disorders) | 2
Conductive deafness (Ear and labyrinth disorders) | 1
Iridocyclitis (Eye disorders) | 1
Papilloedema (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 6
Drug hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 4
Conjunctivitis (Infections and infestations) | 4
Ear infection (Infections and infestations) | 4
Eczema infected (Infections and infestations) | 1
Enterobiasis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Gastritis viral (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Gastroenteritis viral (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 7
Oral fungal infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 6
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Tonsillitis bacterial (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 4
Skin abrasion (Injury, poisoning and procedural complications) | 1
CSF white blood cell count increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 4
Motor developmental delay (Nervous system disorders) | 1
Speech disorder developmental (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hearing aid therapy (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.